CLINICAL TRIAL: NCT07046715
Title: An Open-label, Randomized, Fed, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety After Single-administration of DA-5222 and Co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in Healthy Adult Subjects
Brief Title: Clinical Trial Comparing Single-administration of DA-5222 and Co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in Healthy Adult Subjects in Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5222_BEF_I
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: DA-5222, DA-5222-R1, DA-5222-R2, DA-5222-R3
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5222; Drug: DA-5222-R1; Drug: DA-5222-R2; Drug: DA-5222-R3
- Sequence B (Experimental)
  Interventions: Drug: DA-5222; Drug: DA-5222-R1; Drug: DA-5222-R2; Drug: DA-5222-R3

INTERVENTIONS:
Drug: DA-5222 — single dose administration (DA-5222 one tablet once a day)
Drug: DA-5222-R1 — single dose administration (DA-5222-R1 one tablet once a day)
Drug: DA-5222-R2 — single dose administration (DA-5222-R2 one tablet once a day)
Drug: DA-5222-R3 — single dose administration (DA-5222-R3 one tablet once a day)

SUMMARY:
This study is to compare pharmacokinetics and safety profiles of single-administration of DA-5222 and co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in healthy adult subjects in fed state

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male≥50kg, Female≥45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted
* Subjects with allergy or drug hypersensitivity

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
AUCt | pre-dose~48 hours post-dose
  Area Under the Curve
Cmax | pre-dose~48 hours post-dose
  Maximum Plasma Concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Seoul, Gangseo-gu, South Korea